CLINICAL TRIAL: NCT01633762
Title: Eradication of Gut Microbiota - Effects on Postprandial Gut Hormone Secretion, Glucose Metabolism, Bone Metabolism and Gut Microbiome
Brief Title: Eradication of Gut Microbiota
Acronym: ERA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); Steno Diabetes Center Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristian Hallundbuk Mikkelsen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERA 2012
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes; Obesity; Osteoporosis; Inflammation
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Osteoporosis; Inflammation | interventions — Meropenem; Gentamicins; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- meropenem, gentamicin, vancomycin (Experimental)
  Interventions: Drug: meropenem, gentamicin, vancomycin (together)

INTERVENTIONS:
Drug: meropenem, gentamicin, vancomycin (together) — 4 days antibiotic treatment, per oral, once daily: vancomycin 500 mg (Vancomycin "Hospira"), powder for concentrate; gentamycin 40 mg ("Hexamycin®"), solution; meropenem 500 mg (Meropenem "Hospira"), powder for concentrate; The three drugs are dissolved and combined to a cocktail (with approximately 100 ml of apple juice)

SUMMARY:
The aim of the study is to assess the effect of eradication of gut microbiota on 1) glucose metabolism including postprandial plasma responses of the incretin hormones GIP and GLP-1, insulin, C-peptide and glucagon, 2) metabolomic profiles and resting energy expenditure (REE) 3) appetite, satiety, food intake, gastric emptying and gall bladder emptying, 4) levels of markers of bone formation and resorption as well as serotonin, 5) markers of systemic inflammation, and 6) on the (prospective) composition of bacteria in faeces, blood and saliva. Thus, the overall objective is to provide detailed knowledge on the physiological role of gut microbiota combined with bioinformatic analyses of the functional implications of changes in bacteria composition on the level of both species and phylum.

ELIGIBILITY:
Inclusion Criteria:

* danish caucasian ethnicity
* informed consent
* normal fasting plasma glucose
* normal HbA1c (<6 %)
* normal serum lipids
* normal thyroid function
* normal danish diet
* non-smoking
* normal stool habits

Exclusion Criteria:

* known bone disease
* liver disease (ALAT or ASAT >2 upper normal value)
* kidney disease (serum creatinine >130 μM)
* anaemia
* BMI <18.5 kg/m2 or BMI >25 kg/m2
* known gastrointestinal disease (including prior bariatric surgery,lactose -intolerance, celiac disease, inflammatory bowel disease) or known familial disposition for lactose intolerance, celiac disease, inflammatory bowel disease
* antibiotic treatment within 6 months prior to study including malaria prophylaxis
* medication which cannot be on hold for the study period
* contraindications against/allergy towards the used antibiotics (including prior allergic reactions related to beta-lactam antibiotics, aminoglycosides or vancomycin)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
changes in postprandial GLP-1 secretion | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  plasma level of GLP-1 at baseline and during a 4 hour-meal test

SECONDARY OUTCOMES:
changes in postprandial insulin/c-peptide secretion | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  plasma level of insulin/C-peptide at baseline and during a 4 hour-meal test
changes in postprandial glucose levels | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  plasma level of glucose at baseline and during a 4 hour-meal test
changes in postprandial GLP-2, glucagon, PYY, oxyntomodulin, gastrin, CCK, GIP, leptin, adiponectin and ghrelin secretion | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  plasma levels of GLP-2, glucagon, PYY, oxyntomodulin, gastrin, CCK, GIP, leptin, adiponectin and ghrelin at baseline and during a 4 hour-meal test
changes in markers of bone formation and resorption | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  fasting plasma levels of osteocalcin, P1NP, CTX, 1CTP, sklerostin and serotonin
gut microbiome composition | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  faecal bacterial composition determined from microbiological cultures and deep metagenomic next-generation sequencing of bacterial DNA in feces
changes in markers of systemic inflammation | 0, 4, 42 and 180 days after antibiotic eradication of gut bacteria
  plasma levels of high sensitive CRP, LPBP, TNF-alfa, IL-6 and PAI
changes in glycated hemoglobin (HbA1c) | 42 days after antibiotic eradication of gut bacteria
  plasma level of glycated hemoblobin
changes in body weight | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
changes in basal metabolic rate and respiratory quotient | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  indirect calorimetry measurements (210 minutes postprandial)
changes in gastric emptying | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  1,5 grams of paracetamol will be added to a standardized meal, plasma paracetamol will be measured at baseline and succeeding 4 hours postprandial
changes in gall bladder emptying | 0, 4 and 42 days after antibiotic eradication of gut bacteria
  ultrasonic determination of gall bladder dimensions at baseline and during a 4 hour-meal test (expressed as gall bladder ejection fraction)
appetite, satiety and food intake | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  the impact of eradication on alimentary processes and appetite regulation will be measured using questionnaires and food intake measures
changes in ketone metabolism | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  measurement of fasting plasma beta-hydroxybutyrate level
changes in bile acid deconjugation | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  measurement of feces bile acid (conjugated and deconjugated) concentration to study the effect of gut microbiome presence on bile acid deconjugation
changes in plasma lipid levels | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  fasting plasma levels of triglyceride, VLDL, LDL, HDL, total cholesterol, in addition: measurements of free fatty acids during a 4 hour meal 0, 4 and 42 days after eradication (not on day 8 and 180)
microbiome in blood, urine and saliva | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  measurements on bacteria or bacterial components in blood, urine and saliva to study the effects of gut eradication on blood, urine and saliva microbiome
adverse effects of the used antibiotics | up to 180 days after antibiotic eradication of gut bacteria
  standardized questionaries regarding gastointestinal function are filled out at each study visit (0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria) to detect possible adverse effects of antibiotics. In addition, subjects are given a calendar and informed to write down any symptom or illness during the study period.
changes in metabolomic profile | 0, 4, 8, 42 and 180 days after antibiotic eradication of gut bacteria
  plasma and urine samples for metabolomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kristian H Mikkelsen, MD, Study Director — Diabetes Research Unit, Gentofte Hospital
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Mikkelsen KH, Frost M, Bahl MI, Licht TR, Jensen US, Rosenberg J, Pedersen O, Hansen T, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Effect of Antibiotics on Gut Microbiota, Gut Hormones and Glucose Metabolism. PLoS One. 2015 Nov 12;10(11):e0142352. doi: 10.1371/journal.pone.0142352. eCollection 2015. PMID 26562532